

# STATISTICAL ANALYSIS PLAN

| Study Title: | GENETIC-AF – A <u>Gen</u> otype-Directed Comparative <u>E</u> ffectiveness <u>Trial</u> of Bucindolol and Toprol-XL for Prevention of Symptomatic <u>A</u> trial <u>F</u> ibrillation/Atrial Flutter in Patients with Heart Failure |
|---|---|
| Sponsor: | ARCA biopharma, Inc.<br>11080 CirclePoint Road, Suite 140<br>Westminster, Colorado 80020<br>Phone: 720.940.2100 |
| Study Drug: | Bucindolol hydrochloride (bucindolol) |
| Comparator: | Metoprolol succinate (Toprol-XL, metoprolol) |
| IND No.: | 118,935 |
| Indication: | Atrial Fibrillation |
| Protocol ID: | BUC-CLIN-303 |
| Date: | 15 March 2017 |

Note: The interim analysis methodology is not included in this plan. That methodology can be found in the DSMB Charter and DSMB Statistical Analysis Plan documents.

IND 118,935 

# **TABLE OF CONTENTS**

| 1 | | INITIONS OF ANALYSIS POPULATIONS AND ENDPOINT FOLLOW-UP IODS | 2 |
|---|---|---|---|
| 2 | PAT | TENT CHARACTERISTICS | _ |
| | 2.1 | Screen Failure | |
| | 2.2 | Randomization | 4 |
| | 2.3 | Baseline Characteristics | 4 |
| 2.4 Treatment Exp | | Treatment Exposure and Compliance | 4 |
| | 2.5 | Concomitant Medications | 5 |
| | 2.6 | Metrics for Key Study Procedures | 5 |
| | 2.7 | Final Study Disposition | 6 |
| | 2.8 | Protocol Deviations | 6 |
| 3 | EFF | ICACY ANALYSIS | 6 |
| | 3.1 | General Methodology | 6 |
| | 3.1. | 1 Time-to-Event Analysis Methodology | E |
| | 3.1. | 2 Components of Combined Endpoints | , |
| | 3.1. | 3 Adjudication | / |
| | 3.1. | 4 Core Lab and Transtelephonic Monitoring | 8 |
| | 3.1. | 5 Hospitalization | 8 |
| | 3.1. | 6 Data Collection Cut-off at End of Study | 8 |
| | 3.1. | 7 Missing Data Due to Withdrawal or Loss to Follow-up | 5 |
| | 3.1. | 8 P-value Adjustment for Interim Analysis | 5 |
| | 3.2 | Efficacy Endpoints | 5 |
| | 3.2. | 1 Primary Efficacy Endpoint | 5 |
| | 3.2. | 2 Secondary Efficacy Endpoints | 3 |
| | 3.2. | 3 Tertiary Efficacy Endpoints | 5 |
| 4 | | ETY ANALYSIS18 | - |
| 5 | ME. | ASUREMENTS OF INTEREST AND SUBSTUDIES22 | 2 |

# 1 DEFINITIONS OF ANALYSIS POPULATIONS AND ENDPOINT FOLLOW-UP PERIODS

The efficacy analysis will follow the intent-to-treat (ITT) principle and all patients randomized to study treatment will be included regardless of (1) the success of the treatment titration process and (2) result of electrical cardioversion (ECV) aimed at converting atrial fibrillation (AF) to sinus rhythm (SR). As an additional sensitivity analysis, testing of the primary and secondary endpoints will be repeated on a protocol-compliant subpopulation. Further sensitivity analyses specific to endpoints are described below. The safety analyses will include all patients that received at least one dose of blinded study treatment. The screened population includes any patient who signs informed consent for the study. The screen failure population is a subpopulation of the screened population who are not randomized to study drug for any reason.

Four follow-up periods will be defined for inclusion of each patient's results in endpoint calculations:

- Drug Titration Period: starts on the day of randomized treatment initiation and extends for six weeks after randomization.
- 24-Week Follow-up Period: starts on the day of 1) the first ECG that establishes stable SR (defined in Section 3.2.1), or; 2) the last ECV attempt for patients who fail to convert to stable SR, or; 3) the Week 0 Visit, for patients in AF who do not undergo ECV for any reason. Ends on the day of the Week 24 Visit or the End of Study (EOS) Visit, if patient discontinues prior to Week 24 Visit.
- Total Follow-up Period: starts on the same day as the 24-Week Follow-up Period and extends until the EOS Visit.
- Total Study Period: starts on the day of the Randomization Visit and extends until the EOS Visit.

**Bucindolol HCl** March 15, 2017

# PATIENT CHARACTERISTICS

#### 2.1 **Screen Failure**

Screen failure reasons will be tabulated in order of frequency. These reasons are collected on the eCRF DEMOG form.

#### 2.2 Randomization

Randomized treatment assignment is centralized and in versions 1 and 2 of the protocol was stratified by: 1) HF etiology (ischemic/non-ischemic); 2) LVEF ( $< 0.35 / \ge 0.35$ ) and; 3) type of Medtronic device (Reveal/Non-Reveal/No Device). In protocol version 3 a fourth strata was added: rhythm status at randomization: (SR vs AF). The count of patients randomized by strata within each treatment group will be tabulated by site and overall. The randomization process will be described in full detail.

#### 2.3 **Baseline Characteristics**

The treatment groups will be examined for comparability with respect to demographics, cardiovascular history, AF risk factors, current disease state, HF and AF therapies, physical exam abnormalities, CYP2D6 and  $\alpha_{2C}$  genotyping, vital signs, ECG and laboratory parameters using descriptive statistics. Continuous variables will be analyzed with a mean, standard error, standard deviation, median, minimum, maximum and n=count of results available. Categorical variables will be described with n=count of results available and percentage of study population, with a clear explanation of the denominators provided in footnotes when necessary.

#### 2.4 **Treatment Exposure and Compliance**

The treatment groups will be examined for comparability with respect to the outcome of the titration period (broken down by pre-study beta blocker usage), the attainment of target dose and the days of double blind treatment by dose level and overall. Elapsed days and days of treatment exposure during the four follow-up periods will also be described by treatment group.

Compliance since the previous visit is reported by the sites on the VISREC eCRF form. Overall compliance rates for the 24-Week Follow-up Period and the Total Study Period will be calculated for each patient and compared between the two treatment groups with

 IND 118,935 CONFIDENTIAL descriptive statistics. Note that if a patient discontinues study treatment, compliance is calculated through the date of discontinuation.

#### 2.5 Concomitant Medications

Patients must be receiving optimal anticoagulation therapy for stroke prevention. A tabulation of anticoagulant drug usage by treatment group will be generated. For warfarin users, INR is collected on the LAB eCRF as the following ranges:  $< 1, \ge 1$  and  $< 2, \ge 2$  and  $< 3, \ge 3$  and  $< 4, \ge 4$ . A tabulation of these reported ranges by treatment group will be generated for each of the study visits in which reporting is required.

Reported usage of all concomitant medications during the study will be standardized with preferred name and Anatomical Therapeutic Classification (ATC) using the WHODrug dictionary for tabulation by treatment group.

# 2.6 Metrics for Key Study Procedures

Metrics for the following study procedures and medical interventions will be presented with descriptive statistics by randomized treatment group:

- The cardiac rhythm status of every patient at both the Randomization Visit and at the start of the 24-Week Follow-up Period will be tabulated as follows.
  - Patients in Stable SR at Week 0 who did not require ECV
    - Pts in SR at Randomization
    - Pts in AF at Randomization
  - Patients in Stable SR at Week 0 who did require ECV
    - Pts in SR at Randomization
    - Pts in AF at Randomization
  - Patients in AF/AFL at Week 0
    - Pts in SR at Randomization
    - Pts in AF at Randomization
  - Death/Loss to Follow-up (LTF) prior to Week 0
    - Pts in SR at Randomization
    - Pts in AF at Randomization
- Elapsed days on treatment prior to ECV.
- Outcome of ECV.

- Compliance with procedures for collection of transtelephonic monitoring (TTM) results, and
- Compliance with procedures for collection of Medtronic device results.

# 2.7 Final Study Disposition

The disposition of patients screened and randomized into the study will be tabulated by treatment group and displayed with a flow diagram. This will include the counts of screens, screen failures, re-screens, randomizations, completion of the Week 24 Visit, reasons for permanent discontinuation of study treatment and reasons for discontinuation of study follow-up (broken down by pre/post Week 24 Visit). Note that all patients classified as completing the Week 24 Visit will have all components of the primary and secondary endpoints ascertained through the entire 24-Week Follow-up Period.

#### 2.8 Protocol Deviations

ARCA Clinical Operations maintains an Excel spreadsheet of protocol deviations reported during the study. Each protocol deviation is classified as being Major or Minor, based on its potential impact on clinical results per ARCA SOP CLIN-005. Tabulations and listings of the reported protocol deviations will be provided for both treatment groups.

# 3 EFFICACY ANALYSIS

# 3.1 General Methodology

# 3.1.1 Time-to-Event Analysis Methodology

Time-to-event is calculated as the date of the event minus the date of initiation of efficacy follow-up, with 1 added in order to include both the start date and end date of the interval.

For all endpoints, follow-up will be censored when a patient receives a cardiac transplant, is declared to be permanently lost to follow-up or withdraws consent. The follow-up periods and specific censoring rules are identified in the endpoint descriptions.

These analyses will be a two-tailed comparison of bucindolol and metoprolol, using the log rank statistic with the exact variance calculation stratified by the randomized treatment assignment strata: 1) HF etiology (ischemic/non-ischemic); 2) LVEF ( $< 0.35/ \ge 0.35$ ); 3) type of Medtronic device (Reveal/Non-Reveal/No Device); and 4) rhythm status at randomization:

IND 118,935 

(SR vs AF). Note that patients enrolled under versions 1 and 2 of the protocol were not stratified by rhythm status however their rhythm status is known due to inclusion criteria (all were in AF). The calculations will be performed with the SAS® LIFETEST procedure, with the stratification variables specified in the STRATA statement and the TEST statement used to specify the treatment group comparator and any covariates being examined. Cox's proportional hazards model will be used to calculate estimated hazard ratios and 95% confidence intervals. The calculations will be performed with the SAS PHREG procedure, with the stratification variables specified in the STRATA statement and the treatment group comparator and any covariates being examined specified in the MODEL statement. For the primary endpoint, the appropriateness of assuming proportional hazards will be explored by the graphing of log (-log(survival function)) over follow-up for each treatment group.

Where appropriate, Kaplan-Meier survival curves for bucindolol versus metoprolol will be generated to provide a graphical comparison of the two treatment groups.

Follow-up for the time-to-event endpoints will generally end either at the Week 24 Visit or the EOS Visit for the Total Follow-up Period or Total Study Period endpoints. If the Week 24 Visit falls later than day 180, follow-up will be censored on day 180.

# 3.1.2 Components of Combined Endpoints

This report will contain many endpoints that involve the time to the first occurrence of multiple events, such as AF/AFL onset, mortality or hospitalization. For these endpoints, the count of first events provided by each component will be tabulated. In addition, each component of the combined endpoints will be analyzed separately with a time-to-first-event analysis following the same methodologies used for the combined statistic.

#### 3.1.3 Adjudication

A Clinical Events Classification (CEC) group will adjudicate the primary endpoint, first symptomatic AF/AFL event or death during the 24-Week Follow-up Period. As part of the adjudication process for the primary endpoint, the CEC will also evaluate the secondary endpoint of first AF/AFL event (i.e., symptomatic or asymptomatic). Specifically, the ECGs for the first report of AF/AFL will be reviewed and adjudicated for the presence of AF/AFL regardless of the symptom status. If the first protocol-defined AF/AFL event is not

IND 118,935 

considered a symptomatic AF/AFL event, the triggering process will continue for that patient until the first symptomatic AF/AFL event is identified for the primary endpoint. The CEC over-read of ECG tracings will be used in the calculation of other pertinent study endpoints (such as non-symptomatic AF/AFL within the 24-Week Follow-up Period). More details can be found in the CEC Charter.

# 3.1.4 Core Lab and Transtelephonic Monitoring

In the original study protocol, an Electrophysiology Core Lab (Agility Centralized Research Services) provided a centralized ECG interpretation of the individual ECGs performed at the clinic site and the transtelephonic monitors (TTM) worn by the patients, both during the 24-Week Follow-up Period. In version 4 of the protocol, the collection of these two sources of data was discontinued. The CEC adjudication process was not in production mode at that time point, so it was decided the CEC would perform their own interpretation (over-reads) of the site ECG tracings and not use any of the Core Lab interpretations. Further, the CEC adjudication would make use of available TTM data.

# 3.1.5 Hospitalization

Many of the efficacy endpoints involve hospitalization. Only non-voluntary, overnight hospital admissions will be included in these endpoints; emergency room visits will not be included. Patients in this study will often have scheduled hospital admissions for treatment of their AF and/or HF. Examples include ablation procedures, Tikosyn induction, placement/replacement of implanted devices, and IV drug treatment. These will not be included in the endpoints. The eCRF specifically collects the investigator's assessment of hospitalization causation, which includes assessments of non-CV, CV and HF hospitalizations. In addition to the investigator assessment of causation, the data will be reviewed by the Sponsor via a blinded listing review prior to database lock to confirm which hospitalizations are considered voluntary, overnight admissions.

## 3.1.6 Data Collection Cut-off at End of Study

The protocol states the study will end with approximately 620 randomized patients and accrual of at least 330 primary endpoint events, presuming the sample size and target event counts are not altered due to the Phase 3 interim analysis (see DSMB Charter). At this point, any patients still participating in the 24-Week Follow-up Period will remain on blinded study

IND 118,935 

treatment until they complete the Week 24 Visit. Those patients in the Extension Period will be called in for an EOS Visit.

# 3.1.7 Missing Data Due to Withdrawal or Loss to Follow-up

The rate of withdrawal or loss to follow-up prior to the Week 24 Visit is expected to be low. If a withdrawal or loss to follow-up occurs prior to the Week 24 Visit, all time-to-event endpoints will be censored as of the last completed visit. Note that patients that withdraw from the study will be requested to consent to have their vital status checked via phone calls. If deaths are detected by this procedure the date of death will be incorporated into the efficacy and safety datasets and analyses.

# 3.1.8 P-value Adjustment for Interim Analysis

The goals and operational details for the interim efficacy analysis and ongoing safety monitoring can be found in the DSMB Charter and the DSMB SAP.

At the end of Phase 3, the alpha level for the primary endpoint will be reduced to 0.04989 to adjust for the Phase 2B ( $\alpha = 0.00001$ ) and Phase 3 ( $\alpha = 0.0001$ ) interim analyses.

# 3.2 Efficacy Endpoints

# 3.2.1 Primary Efficacy Endpoint

The primary endpoint is elapsed time-to-first-event of symptomatic AF/AFL or all-cause mortality (ACM) during the 24-Week Follow-up Period. This is a time-to-event endpoint censored at the end of the 24-Week Follow-up Period. The identification of first event of symptomatic AF/AFL or death is provided by the CEC. The CEC does not distinguish between the presence of AF or AFL so a component analysis will not be possible.

The following definitions apply to this endpoint:

- Stable SR on study drug is defined as any of the following:
  - SR confirmed  $\geq 1$  hour after ECV.
  - SR confirmed  $\geq 1$  hour after spontaneous conversion from AF/AFL.
  - SR confirmed  $\geq 1$  hour at the Week 0 Visit for patients randomized in SR.
- An AF/AFL event is defined as AF or AFL observed on two consecutive measures separated by at least 10 minutes as assessed by ECG/TTM.

 A symptomatic AF/AFL event is defined as an AF/AFL event that is associated with a clinically relevant change in patient-reported symptoms, as determined by the CEC examination of blinded data.

The CEC charter and associated documents describe the "triggers" that are established to identify events for their consideration and the data sources to be used in their adjudication proceedings. The charter also describes their approach for identifying an AF event as symptomatic and for identifying the onset date and time of the event since that is needed for this time-to-event endpoint. Note that version 3 of the protocol involved a comprehensive change to the symptoms collected, with 6 of the original 8 symptoms having their descriptions modified and 2 new symptoms being added. Also the symptom characteristics were clarified with addition of a 'frequency' field to the collection form. All of these changes were made to give the CEC more specific information to support their identifying symptoms that were new or worsened in association with AF onset. Since these changes were implemented after only 12 patients were randomized (2% of the planned 620) and the identification of overall symptom onset/worsening is an adjudicated decision, no modification of analysis methodology is planned.

AF/AFL will be assessed at scheduled and unscheduled clinic visits via 12-lead ECG. Patients will be queried at the time of each ECG assessment to determine if they have experienced any change in symptoms that could be potentially related to AF.

The vast majority of patients will either be in SR or successfully convert from AF to SR after one or two ECV procedures around three weeks after they begin randomized treatment. However, there are several scenarios that depart from this norm and the methodology for establishing the start of efficacy follow-up and censoring for the primary endpoint is described below:

- 1. Spontaneous conversion to stable SR prior to the planned cardioversion. For these patients, the day of the first ECG assessment that meets the definition of stable SR, as defined above, will be designated as Day 1 of the 24-Week Follow-up Period.
- 2. Failure to attain stable SR because the ECV procedure was not performed due to drop out or any reason other than those described below. These patients will be included in the analysis as censored on Day 1 of the 24-Week Follow-up Period.

IND 118,935 

- 3. Failure to attain stable SR, either spontaneously or following ECV. These patients will be included in the endpoint calculation as experiencing the event on Day 1 of the 24-Week Follow-up Period.
- 4. Deaths occurring after randomization and prior to conversion to stable SR will be counted as events on Day 1 of the 24-Week Follow-up Period.
- 5. Patients with AF/AFL stopped at the Week 0 Visit by any means other than ECV will be censored on Day 1 of the 24-Week Follow-up Period. An example is the performance of AV nodal ablation at the Week 0 Visit.

The primary endpoint analysis will also be performed within the following prospectively identified subgroups based on pathophysiological or clinical importance:

- 1) Started the 24-Week Follow-up Period in SR vs AF
- 2) LVEF strata at randomization: ≤0.35 vs. >35
- 3) Gender
- 4) Ischemic etiology vs. nonischemic
- 5) Age above/below median
- 6) Duration of AF diagnosis above and below median.
- 7) Baseline norepinephrine above and below median
- 8) Baseline NT-proBNP
- 9)  $\alpha_{2C}$  AR polymorphisms (i.e., Del carriers vs.  $\alpha_{2C}$  wild type homozygotes).

In exploratory analyses, the following covariates will be included as potentially relevant explanatory variables in the Cox regression models:

- 1. Initial study treatment dose level.
- 2. Baseline NYHA Class.
- 3. Gender.
- 4. Race.
- 5. Age.
- 6. Baseline serum creatinine.
- 7. Baseline norepinephrine level.
- 8. Baseline heart rate.

- 9. Baseline systolic blood pressure.
- 10. History of diabetes.
- 11. Duration of AF diagnosis.
- 12. Previous amiodarone use (both historical and stopped just prior to randomization).
- 13. Ablation procedure prior to study.
- 14. Therapeutic device type: CRT, ICD, single ventricular lead pacemaker.
- 15. For the subset of patients in AF at baseline, type of rhythm abnormality: (paroxysmal AF or persistent AF).
- 16. For the subset of patients in SR at baseline: the time since last attaining SR, the type of previous rhythm abnormality, and the intervention that ended the previous AF episode.
- 17. Elapsed days of treatment from randomization date to start of the 24-Week Follow-up Period.
- 18. CYP2D6 metabolizer status.
- 19.  $\alpha_{2C}$  AR polymorphisms (i.e., Del carriers vs.  $\alpha_{2C}$  wild type homozygotes).
- 20. Country in which clinic site is located.
- 21. Other clinically significant AF risk factors.

# Additional exploratory analyses will include the following:

- A qualitative analysis of the symptoms associated with the primary endpoint events. The symptoms will be classified as arrhythmia-related (palpitations or lightheadedness/dizziness) HF-related (fatigue or tiredness, weakness or problems exercise, weight gain or swelling of both legs and/or feet), or both.
- For patients with primary endpoint events of symptomatic AF/AFL, how many had prior events of asymptomatic AF/AF that progressed into symptomatic.

# The following sensitivity analyses will be performed:

- A subpopulation analysis including only those patients beginning the 24-Week Follow-up Period in SR.
- In the per-protocol analysis, endpoint events and deaths that occur more than 30 days after permanent discontinuation of study treatment are omitted.

IND 118,935 

- All Week 24 Visits included (ie no exclusion of events observed at Week 24 Visits after day 180).
- Patients that have not previously reverted to AF/AFL that withdraw or are lost to follow-up prior to the Week 24 Visit, will be assigned an AF/AFL event at the first missed clinic visit or scheduled TTM.
- Patients that withdraw or are lost to follow-up prior to the Week 24 Visit are omitted from the analysis.

# 3.2.2 Secondary Efficacy Endpoints

The following endpoints will be tested for superiority of bucindolol benefit relative to metoprolol by fixed sequence provided that bucindolol is found to be significantly superior in the primary endpoint. The time-to-event endpoint methodology described in Sections 3.1.1 and 3.2.1 for events involving AF/AFL recurrence will be used unless otherwise noted:

• Time-to-first-event of AF/AFL (i.e., symptomatic or asymptomatic) or ACM during the 24-Week Follow-up Period.

# Supportive Analyses:

- Events accrued during the Total Follow-up Period.
- For patients with events based on symptomatic AFL, the rate of patients subsequently progressing to AF. Also for these patients, the elapsed time from symptomatic AFL to AF.

## Data Source:

- ECG (over-read by CEC for first 24 weeks)
- TTM (first 24 weeks only)
- Proportion of patients with VT, VF, or symptomatic supraventricular tachycardia (SVT) during the 24-Week Follow-up Period. Includes VF and symptomatic SVT events of any duration, VT events ≥ 15 seconds, and VT events that result in appropriate firing of an ICD. It will be tested with a Cochran-Mantel-Haenszel statistic to control for the four stratification variables.

IND 118,935 

# Supportive Analyses:

- Events accrued during the Total Follow-up Period.

## Data Source:

- The CVEVENT eCRF form is the source of all components of these compound endpoints.
- Total all-cause hospitalization days per patient during the Total Study Period. The count of hospitalization days will be normalized for the total number of days of follow-up prior to testing with the Wilcoxon Rank Sum statistic.

# Supportive Analyses:

- Number of heart failure hospitalization days per patient.
- All-cause hospitalization days through first recurrence of AF/AFL versus days
  after recurrence, normalized for days of follow-up within each period. The
  comparison will take place within treatment group and across treatment.
- All-cause hospitalization days for patients with ventricular rate control (VRR)
   control compared to those without VRR control. The comparison will take
   place within treatment group and across treatment.

#### Data Source:

- The HOSP eCRF form provides the number of hospitalization days and the reason for hospitalization.
- The ECG and AE eCRF will be used to identify the patients in AF with VRR control at the end of the study.
- Time-to-first-event of AF/AFL (i.e., symptomatic or asymptomatic), HF hospitalization (as assessed by the Investigator), or ACM during the Total Follow-up Period. As in the primary endpoint, any incidence of ACM prior to start of the 24-Week Follow-up Period will be analyzed as an event on Day 1. Hospitalization prior to Week 0 are not included, but those are included in the safety analyses.

# Supportive Analyses:

IND 118,935 

- Events accrued during the 24-Week Follow-up Period.
- Combinations of each component ((i.e., AF/AFL+ACM, AF/AFL+HFH, HFH+ACM).

#### Data Source:

- ECG (over-read by CEC for first 24 weeks), HOSP and DEATH eCRF forms.
- TTM (first 24 weeks only).
- Proportion of patients with adequate ventricular rate control (VRR) in the setting of AF/AFL. Adequate VRR in setting of AF/AFL is defined as follows: 1) the presence of AF or AFL; 2) a VRR between 40 and 80 beats per minute (bpm) at rest; and 3) the absence of symptoms associated with bradycardia. Thus this is a subset analysis only involving patients with AF/AFL recurrence. The endpoint is evaluated for the last tracing demonstrating AF/AFL during the 24-Week Follow-up Period prior to intervention (eg: ablation, ECV, initiation of anti-arrhythmic drugs). Will be tested with a Cochran-Mantel-Haenszel statistic to control for the four stratification variables.

## Supportive Analyses:

 Evaluated for the last tracing demonstrating AF/AFL when the patient is still on study treatment during the 24-Week Follow-up Period.

#### Data Source:

- ECG and AE eCRF form (for symptomatic bradycardia).

# 3.2.3 Tertiary Efficacy Endpoints

The following endpoints will be tested for superiority of bucindolol benefit relative to metoprolol. The time-to-event endpoint methodology described in Sections 3.1.1 and 3.2.1 for events involving AF/AFL recurrence will be used unless otherwise noted:

Time-to-first-event of VT/VF or ACM during the Total Follow-up Period. Includes
VF events of any duration, VT events of ≥ 15 seconds, and VT events that result in
appropriate firing of an ICD.

IND 118,935 

# Supportive Analyses:

- Events accrued during the 24-Week Follow-up Period.

## Data Source:

- CVEVENT and DEATH eCRF forms.
- Time-to-first-event of AF/AFL (i.e., symptomatic or asymptomatic), CV-related hospitalization (as assessed by the Investigator), or ACM during the Total Study Follow-up Period.

# Supportive Analyses:

- Events accrued during the 24-Week Follow-up Period.
- Combinations of each component (i.e., AF/AFL+ACM, AF/AFL+CVH, CVH+ACM).

#### Data Source:

- ECG (over-read by CEC during the 24-Week Follow-up Period), HOSP and DEATH eCRF forms.
- TTM (24-Week Follow-up Period).
- Proportion of patients with stroke or systemic embolism during the Total Follow-up Period. Stroke is defined as a focal neurologic deficit from a non-traumatic ischemic, hemorrhagic, or uncertain cause lasting at least 24 hours (as assessed by the Investigator). Tested with a Cochran-Mantel-Haenszel statistic to control for the four stratification variables.

#### Data Source:

- CVEVENT eCRF form.
- Proportion of patients randomized with AF/AFL who convert to stable SR
  (spontaneous or post-ECV) and enter the 24-Week Follow-up Period. Tested with a
  Cochran-Mantel-Haenszel statistic to control for the four stratification variables.

Supportive Analyses:

Subset of patients with spontaneous conversion.

#### Data Source:

- FUSTART eCRF form.
- Total number of ECV procedures per patient during the Total Study Period. This count will be normalized for the total number of days of follow-up prior to testing with the Wilcoxon Rank Sum statistic.

#### Data Source:

- ECV eCRF form.
- Proportion of patients at Week 24 Visit who are receiving study drug and have not had an AF/AFL event. Tested with a Cochran-Mantel-Haenszel statistic to control for the four stratification variables.

#### Data Source:

- ECG (over-read by CEC), DRUGLOG and EOT eCRF forms.
- TTM (24-Week Follow-up Period).
- Change in NT-proBNP, assessed relative to baseline (Randomization Visit). Change
  from baseline will be tested for greater reduction in the bucindolol treatment group
  with the Wilcoxon Rank Sum test because of the expected lack of normality of this
  measure.

#### Data source:

- LabCorp vendor dataset.
- Change in norepinephrine, assessed relative to baseline (Randomization Visit).
   Change from baseline will be tested for greater reduction in the bucindolol treatment group with the Wilcoxon Rank Sum test because of the expected lack of normality of this measure.

#### Data source:

LabCorp vendor dataset.

• The EQ-5D questionnaire has 5 dimensions (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and each is self-rated by the patient as no problems, some problems, or severe problems. The results for each dimension will be analyzed individually at both time points. The change from randomization to each visit will be categorized as improved or no change/worsened and the proportions of these categories in both treatment groups will be tabulated with a 2 by 2 table. The bucindolol treatment group will be tested for superior response using a Cochran-Mantel-Haenszel statistic to control for the four stratification variables.

Data source:

- EQ-5D eCRF form.
- Pharmacoeconomic modeling of healthcare utilization. Details of this analysis will be prespecified in a separate analysis plan.

# 4 SAFETY ANALYSIS

The following four periods are established for analysis of safety endpoints:

- 24-Week On-Drug Period: starts at day of randomization and extends to latest visit attended through Week 24 Visit. For patients that discontinue treatment early, data collected through 30 days after the final dose of study treatment are included.
- 24-Week On-Study Period: starts at day of randomization and extends to latest visit
  attended through Week 24 Visit. For patients that discontinue the study prior to
  Week 24, data collected through 30 days after the final study visit are included.
  Study treatment status is not considered for data inclusion.
- Total Study On-Drug Period: starts at day of randomization and extends through 30 days after the final dose of study treatment.
- Total Study On-Study Period: starts at day of randomization and extends through 30 days after final clinic visit attended. Study treatment status is not considered for data inclusion.

Analysis of SAEs will be performed for all four timeframes. For the other safety endpoints, the 24-Week On-Study and Total Study On-Study Periods will be used. If treatment group

IND 118,935 

imbalances are observed for an endpoint, it will be further analyzed with the other data inclusion timeframes.

The results for the following safety endpoints will be compared with descriptive statistics between the treatment groups for all patients receiving study treatment. Results collected from first dose of study drug to 30 days after the last dose for each patient will be included in the assessments of safety. Results specific to scheduled visits will be included in the by-visit analyses if they were collected within  $a \pm 7$ -day window for the prescribed visit study day.

• Incidence of ACM during the Total Study Period.

Supportive Analyses:

 The association of VRR control with mortality will be examined using the final heart rate measurement available for each patient (comparisons will be within the treatment groups).

## Data Source:

- DEATH eCRF form.
- Incidence of ACM, CV-related hospitalization (as assessed by the Investigator), or withdrawal of study drug due to an AE during the Drug Titration Period.
   Data source:
  - DEATH, HOSP, EOS and AE eCRF forms.
- Incidence of symptomatic heart block during the Total Study Period. Symptomatic Heart Block is defined as the first of any of the following: 1) 3rd degree heart block (complete heart block); 2) any 2nd degree heart block with the presence of symptoms attributable to, and temporally correlated with the occurrence of heart block which include any of the following: Near-fainting or fainting (syncope) / Dizziness; Weakness or Fatigue; Shortness of breath; Chest pain; or 3) 2nd or 3rd degree heart block requiring implantation of a permanent pacemaker (with or without defibrillator).

#### Data source:

- CVEVENT and AE eCRF forms.

IND 118,935 

 Overall incidence and severity of treatment-emergent AEs/SAEs over time during the Total Study Period. Also events associated with device implantation. The events will have standardized MedDRA preferred terms and System Organ Classes assigned to them for tabulation.

# Supportive analyses:

- Incidence of AEs leading to reduction, interruption or permanent discontinuation of study treatment.
- Incidence of AEs associated with device implantation.
- Incidence of AEs by CYP2D6 metabolizer status.
- Incidence of AEs by  $\alpha$ 2C AR polymorphisms.

#### Data source:

- AE eCRF form.
- Incidence of neoplasm-related AEs during the Total Study Period. The AEs of special interest will be tabulated according to the following characteristics.
  - Development of treatment-emergent neoplastic conditions.
  - Progression or worsening of pre-study neoplastic conditions.
  - Progression or worsening of treatment-emergent neoplastic conditions.

#### Data source:

- AE, NEOPLHX and NEOPLAS eCRF forms.
- Clinical Chemistry and Hematology.
  - Visit collection: screen, start of follow-up Week 0 (protocol versions 1 and 2),
     Week 4 (protocol versions 3 and 4), Week 12 (protocol versions 3 and 4),
     Week 24, every 24 weeks during extension, end of treatment and end of study.
     Screen results will serve as the pre-treatment baseline.
  - Change from baseline to each planned study visit of collection will be calculated and analyzed with descriptive statistics.

IND 118,935 

- The numbers and percentages of patients with values exceeding the bounds of normal ranges will be tabulated for scheduled visits.
- The numbers and percentages of patients with values exceeding the panic bounds each visit.

#### Data source:

- LabCorp vendor-supplied dataset.
- ECG quantitative parameters.
  - Measured at every visit. Randomization Visit measurement prior to first dose will serve as the baseline. Will be analyzed at Week 0, 4, 12 and 24 visits as well as end of treatment and end of study.
  - Change from baseline to each analysis visit will be calculated and analyzed with descriptive statistics.
  - The numbers and percentages of patients with QTc increase from baseline exceeding 60 ms at any time point during the study.

#### Data source:

- ECG eCRF form.
- Vital signs and weight (data source: VITALS eCRF form).
  - Measured at every in-clinic visit. Randomization Visit measurement prior to first dose will serve as the baseline. Will be analyzed at Week 0, 4, 12 and 24 visits as well as end of treatment and end of study.
  - Change from baseline to each analysis visit will be calculated and analyzed with descriptive statistics.

#### Data source:

- VITALS eCRF form.
- Proportion of patients attaining target study drug dose during the Drug Titration
   Period. Will be calculated for all patients, those receiving β-blocker therapy prior to randomization and those not previously receiving β-blocker therapy.

IND 118,935 

#### Data Sources:

VISREC and DRUGLOG eCRF forms.

# 5 MEASUREMENTS OF INTEREST AND SUBSTUDIES

• AF Burden (AFB) Substudy.

In this optional substudy, AFB, defined as the amount of time per day that a patient is in AF/AFL, is measured by implanted Medtronic devices, including cardiac monitors, pacemakers, cardioverter-defibrillators, and cardiac resynchronization therapy. These devices also measure VRR during periods of AF. Approximately 50% of the study participants are expected to participate in the AFB substudy.

The distribution of device types will be presented by treatment group, by patient baseline characteristics, by disease severity, by treatment exposure prior to device implantation and elapsed days to start of the 24-Week Follow-up Period. AFB will be presented as hours/day in graphical displays for each patient with the dates of randomization and initial ECV and other interventions annotated.

The treatment efficacy endpoint will be the time to first device-detected event or ACM, with an event defined as at least 6 hours of AFB in a single day. This endpoint will be analyzed through the Week 24 Visit with the same methodology used for the study primary endpoint. Patients with no AFB data available after the start of the 24-Week Follow-up Period will be excluded. Patients with an implanted therapeutic device that produces paced rhythm which confounds the measurement of AFB will also be excluded.

#### Supportive Analyses:

- Time to device detected AF/AFL event during the Total Follow-up Period.
- The proportion of patients with VRR on the last day demonstrating AF/AFL during the 24-Week Follow-up Period. Will be tested using a Cochran-Mantel-Haenszel statistic to control for the four stratification variables.
- The percent of follow-up days in AFB, calculated as the number of days with
   AFB of at least six hours divided by the total number of days in the 24-Week

Follow-up Period. Statistical testing will be performed with the Wilcoxon Rank Sum Statistic. A sensitivity analysis will be performed on the subset of patients beginning the 24-Week Follow-up Period in SR.

## Data Sources:

- Medtronic vendor-supplied dataset.
- DNA Bank, with collection at time of screening, for patients who agree to participate in the substudy. No analysis of these data have been pre-planned.
- Sparse sampling of bucindolol hydrochloride plasma concentrations for population pharmacokinetic analysis. The analysis plan for the substudy will be prepared separately prior to unblinding.

IND 118,935 